CLINICAL TRIAL: NCT00210860
Title: An Open-label Study of the Safety and Efficacy of Topiramate for Migraine Prophylaxis: Extension Study to CAPSS-277
Brief Title: An Open Label Extension of a Study Comparing Topiramate and Amitriptyline in Migraine Prevention.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR004669
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: chronic; headache; prevention; Migraine
MeSH Terms: conditions — Migraine Disorders; Bronchiolitis Obliterans Syndrome; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the long-term safety and effectiveness of topiramate for the prevention of migraine headaches in adults. Topiramate has been approved to prevent migraine headaches in adults.

DETAILED DESCRIPTION:
Migraine headaches can be disabling and can interfere with work and a person's quality of life. Preventing these headaches before they start is the best option. Topiramate, an anti-seizure medication, has been shown to help prevent migraine headaches from occurring. This is an open-label study that is an extension of a previous study (CAPSS-277) comparing topiramate and amitriptyline in migraine prevention. It includes patients who completed the previous study and elected to enter open label treatment with topiramate. The study will involve a 4-week Blinded Transition Phase during which patients will be titrated up to a daily topiramate dose of 100 milligrams (or the maximum tolerated dose, whichever is less). Then there will be a 12-week Open-Label Maintenance Phase during which the topiramate dose may be adjusted according to effectiveness and tolerance, but not to exceed a daily dose of 400 milligrams. While on topiramate, patients will record daily entries in their headache records. Patients will be asked questions to help assess their quality of life. Patients will also have physical examinations and laboratory tests performed during the study. The objective of this study is to evaluate the long-term safety and effectiveness of topiramate for the prevention of migraine headaches.

Topiramate oral tablets, 25 milligrams per tablet, will be given in the morning and evening to a dose not to exceed 400 milligrams per day or to the maximum tolerated dose, whichever is less

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura
* Successfully finished CAPSS-277 study
* In generally good health
* Able to take medicine orally
* If female, using birth control

Exclusion Criteria:

* Not having a more painful condition than the headache pain
* Cannot be taking any other medications not allowed by the study
* Abnormal liver tests
* Not compliant with study medication during the CAPSS-277 study
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2004-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Patient diary: number, duration, severity of headaches, symptoms, other medications used; QOL: Migraine Disability Assessment, Migraine-Specific Quality of Life, Quality of Life Enjoyment & Satisfaction Questionnaire-Short Form, Weight Satisfaction Scale

SECONDARY OUTCOMES:
Adverse event reports; physical examinations; vital signs; electrocardiogram; laboratory tests for safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label Study of the Safety and Efficacy of Topiramate for Migraine Prophylaxis: Extension Study to CAPSS-277 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=618&filename=CR004669_CSR.pdf